CLINICAL TRIAL: NCT02778997
Title: Prospective Shunt Complication Study (Pro-ShuCS)
Brief Title: Prospective Shunt Complication Study
Acronym: ShuCS
Status: Suspended | Type: Observational
Why Stopped: Responsible investigator left the team. Suspended until replacement is found.
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00174
Record Dates: First submitted 2016-04-25; First posted 2016-05-20 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Shunt; Complications, Ventricular (Communicating)
Keywords: Shunt; CSF; Dysfunction; Complication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: CSF Shunt treatment for hydrocephalus — State after CSF shunt implantation

SUMMARY:
Complications in patients with cerebrospinal fluid (CSF) shunts are common. Thus, these patients are frequently admitted for suspicion of a shunt dysfunction (SD). However, the symptoms of a SD are often unspecific and the required diagnostics are time consuming, expensive, invasive and may involve radiation exposure. In a prospective observational study it is planned to find out, how often a suspected shunt dysfunction is found, which kinds of shunt dysfunction are seen and if there is a correlation between the shunt dysfunctions and the age of the shunt. Furthermore, it is intended to find out, if there are symptom-patterns specific for certain shunt dysfunctions.

DETAILED DESCRIPTION:
All patients who are admitted for suspected shunt-dysfunction will be included. Patient data, detailed data about the shunt, patient's symptoms and all findings will be recorded in the CRF. After 4-8 weeks all patients will be followed-up to add missing data and correct initial findings with the benefit of a retrospective view. After 2 years, data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* State after implantation of a CSF shunt

Exclusion Criteria:

* refusion participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with CSF shunt
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Confirmation of Shunt Dysfunction (yes/no) | 4-8 weeks after first presentation
  The correctness of the suspected diagnosis of a shunt dysfunction
Kind of Shunt Dysfunction (infection/disruption/kinking/obstruction/others) | 4-8 weeks after first presentation
  In case of a confirmed shunt dysfunction, the kind of dysfunction is recorded
Alternate Diagnosis (multiple diagnoses possible) | 4-8 weeks after first presentation
  If the suspected diagnosis of a shunt dysfunction is not approved, the alternate diagnosis leading to the patient's symptoms is recorded. Every possible medical disorder might lead to presentation of the patient. Thus, no catalogue of possible diagnoses is given.
Time Span after Shunt Implantation (months) | 4-8 weeks after first presentation
  Certain kinds of shunt dysfunctions seem to appear at a certain "age" of a shunt. The time after implantation/last revision of the shunt is recorded. The age of the shunt / time span after first implantation is measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Regli, MD, Study Director — Zurich University Hospital, Dept. of Neurosurgery; Lennart H Stieglitz, MD, Principal Investigator — Zurich University Hospital, Dept. of Neurosurgery
Locations (2):
- Switzerland (2):
  - Dept. of Neurosurgery, Zurich University Hospital, Zurich
  - Zurich University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: No